CLINICAL TRIAL: NCT01647906
Title: A Prospective, Single Arm, Multicenter, Observational Assessment of the Long Term Safety and Efficacy of Solesta® Injectable Bulking Agent for the Treatment of Fecal Incontinence (SoFI)
Brief Title: Long Term Safety and Efficacy of Solesta® Injectable Bulking Agent for the Treatment of Fecal Incontinence (SoFI)
Acronym: SoFI
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL SLP001
Record Dates: First submitted 2012-06-27; First posted 2012-07-24 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to evaluate the safety and effectiveness of the Solesta Injectable Bulking Agent in the treatment of fecal incontinence through 3 years in a real world setting.

DETAILED DESCRIPTION:
This observational study is to evaluate the safety and effectiveness of the Solesta Injectable Bulking Agent in the treatment of fecal incontinence through 3 years in a real world setting.

ELIGIBILITY:
Inclusion Criteria: A patient will be eligible for study participation if he/she meets the following criteria:

* Able to fluently speak and understand the language in which the study is being conducted and able to provide meaningful written informed consent for the study.
* Have FI, have failed conservative therapy (e.g., diet, fiber therapy, medications that treat diarrhea), and are scheduled to receive Solesta treatment.
* Females must be of non-childbearing potential; or females of childbearing (reproductive) potential must agree to use an acceptable method of contraception for at least the first 6 months of study participation and have a negative urine pregnancy test at Visit 1 (Screening/Baseline) and immediately prior to receiving initial Solesta treatment. Women who are surgically sterile or those who are post menopausal for at least 2 years prior to entering the study are not considered to be of childbearing potential.
* Willing to return to the study facility for the post treatment evaluation.

Exclusion Criteria: A patient will be excluded from the study if he/she meets any of the following criteria:

* Is currently pregnant, breastfeeding, or is planning to become pregnant over the course of the study.
* Has an active inflammatory bowel disease.
* Has an immunodeficiency disorder or ongoing immunosuppressive therapy.
* Has received previous radiation treatment to the pelvic area.
* Has significant mucosal or full thickness rectal prolapse.
* Has active anorectal conditions including: abscess, fissures, sepsis, bleeding, proctitis, or other infections.
* Has anorectal atresia, tumors, stenosis or malformation.
* Has a rectocele.
* Has rectal varices.
* Has presence of existing implant including Solesta, artificial bowel sphincter, or sacral nerve stimulator (activated or inactivated).
* Has an allergy to hyaluronic acid (HA) based products.
* Has an anastomosis to the rectum or anus within 10 cm of the dentate line.
* Has an unstable condition (e.g., psychiatric disorder, a recent history of substance abuse) or otherwise thought to be unreliable or incapable of complying with the requirements of the post-approval study protocol.
* Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study.
* Has undergone sphincteroplasty, graciloplasty, or other surgical interventions (without the use of an implanted device) for treatment of fecal incontinence within 12 months of enrollment.
* Has any bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Fecal Incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Freedom from fecal incontinence reintervention | Through 36 months after the last Solesta treatment
  The primary effectiveness endpoint is freedom from Fecal Incontinence Reintervention. Patients will be evaluated at 3, 6, 12, 24, and 36 months after the last Solesta treatment for the occurrence (or lack of occurrence) of Fecal Incontinence Reintervention. Fecal Incontinence Reintervention includes Fecal Incontinence treatment of sphincteroplasty, implantation of artificial bowel sphincter, retreatment with Solesta, graciloplasty, sacral nerve stimulation (SNS) or other surgical interventions that occur more than 3 months after the last primary Solesta treatment.

SECONDARY OUTCOMES:
Fecal Incontinence Quality of Life (FIQL) | Assessed at baseline, 3, 6, 12, and 36 months after last Solesta treatment.
  The effectiveness endpoint of Fecal Incontinence Quality of Life using the Rockwood instrument will be assessed at baseline, 3, 6, 12, and 36 months after last Solesta treatment. Patients will fill out a questionnaire at screening visit and at follow up visits. The Fecal Incontinence Quality of Life instrument is a questionnaire completed by patients that assesses the impact of quality of life as it relates to Lifestyle, Coping/Behavior, Depression/Self perception and Embarrassment. The FIQL instrument consists of a total of 29 questions.
Cleveland Clinic Florida Fecal Incontinence Score (CCFIS) | Assessed at baseline,3, 6, 12, and 36 months after last Solesta treatment
  The effectiveness endpoint of CCFIS will be assessed at baseline, 6, 12, and 36 months after last Solesta treatment. The investigator will calculate the CCFIS based on a patient interview. The CCFIS is a summed score of 5 individual parameters (i.e., frequency of incontinence to gas, liquid, solid, of need to wear pad, and of lifestyle changes).
Global Perceived Effect Score | Assessed at 6, 12 and 36 months after last Solesta treatment
  The effectiveness endpoint of Global Perceived Effect Score will be assessed at 6, 12 and 36 months after last Solesta treatment. Global perceived effect is a subjective score and reflects the patient perception of their degree of FI after treatment compared to the period before treatment and ranges from 1-7 points.
Time to Fecal Incontinence Reintervention | Assessed from 6 to 36 months after last Solesta treatment
  For patients who undergo Fecal Incontinence Reintervention the effectiveness endpoint of Time to Fecal Incontinence Reintervention will be measured from the date of last treatment with Solesta to the date of first Fecal Incontinence Reintervention. Fecal incontinence reinterventions will include any of the following FI treatments: sphincteroplasty, implantation of artificial bowel sphincter, retreatment with Solesta, graciloplasty, SNS or other surgical interventions.
Anatomic stability of the Solesta | Assessed at time of Solesta treatment and again at 6 and 36 months after the last Solesta treatment.
  Assess the relative anatomic stability of the Solesta Injectable Bulking Agent in a subpopulation of patients enrolled at 3-4 sites as assessed by transrectal ultrasound. Solesta will be assessed by comparing anatomical positioning of the Solesta implant, as determined by transrectal ultrasound at Visit 3a (for patients who did not receive a second Solesta treatment) or Visit 3b (for patients who received a second Solesta treatment at Visit 3a) to positioning at 6 and 36 months after the last Solesta treatment.
Occurrence of any peri-injection device related infectious adverse events. | Assessed from time of injection up to 2 weeks after Solesta treatment
  A secondary safety endpoint will be the occurrence of peri-injection device related infectious Adverse Events for patients treated with or without prophylactic antibiotics (as decided by treating physician) prior to injection.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Mayo Clinic, Scottsdale, Arizona
  - Colon and Rectal Medical Services, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Galliano Private Practice, Port Charlotte, Florida
  - USF Health, Tampa, Florida
  - North Pinellas Surgical Institute, Tarpon Springs, Florida
  - Cleveland Clinic Florida Health, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Regents Research Institute, Augusta, Georgia
  - The Iowa Clinic, Des Moines, Iowa
  - Colon and Rectal Surgery Associates, Ltd., Minneapolis, Minnesota
  - Colon and Rectal Surgery, LLC, Omaha, Nebraska
  - North Shore Long Island Jewish Health Systems, Huntington, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Cleveland Clinic Foundation Digestive Disease Institute, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Colon and Rectal Research Foundation, Allentown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont

REFERENCES:
- [Derived] Quiroz LH, Galliano DE Jr, da Silva G, Carmichael JC, Pan LC, Bromley ER, Hinahara JG, Goss TF. Efficacy and Safety of a Nonanimal Stabilized Hyaluronic Acid/Dextranomer in Improving Fecal Incontinence: A Prospective, Single-Arm, Multicenter, Clinical Study With 36-Month Follow-up. Dis Colon Rectum. 2023 Feb 1;66(2):278-287. doi: 10.1097/DCR.0000000000002348. Epub 2023 Jan 4. PMID 35001051